CLINICAL TRIAL: NCT01200641
Title: Evaluation of Anxiolysis and Pain Associated With Retrobulbar Eye Block for Cataract Surgery : Melatonin Versus Gabapentin ( A Randomized, Double-blind, Placebo-controlled Study)
Brief Title: Evaluation of Anxiolysis and Pain Associated With Retrobulbar Eye Block for Cataract Surgery : Melatonin Versus Gabapentin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Qazvin University Of Medical Sciences, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12610000727044
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Anxiety; Pain
Keywords: melatonin; gabapentin; anxiety; pain; retrobulbar block
MeSH Terms: conditions — Anxiety Disorders; Pain | interventions — Melatonin; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- melatonin (Active Comparator): ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Interventions: Drug: Melatonin
- gabapentin (Active Comparator): ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator): ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Melatonin — ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Arms: melatonin
Drug: Gabapentin — ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Arms: gabapentin
Drug: placebo — ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6
  mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) orally 90 minutes before retrobulbar injection( for all of three groups).
  Arms: placebo

SUMMARY:
Principle goals of sedation for eye surgery are to provide patient comfort and to allow the patient to stay calm during both retrobulbar injection and surgery. Insufficient sedation may not prevent the patient from moving during retrobulbar injection, whereas very deep sedation may result in respiratory complications during surgery .The investigators compared the effect of melatonin and gabapentin on the hemodynamic parameters, sedation ,anxiety, and pain and satisfaction profile in cataract surgery. After approval by the Hospital Evaluation Committee of Scientific Studies for ethical purpose and written informed consent, ninety patients scheduled for cataract surgery by phacoemulsification were randomly allocated to three study groups to receive melatonin 6 mg (Group M, n = 30) , gabapentin 600mg(GroupG, n = 30)or placebo(GroupP, n=30) 90 minutes before retrobulbar injection. . Hemodynamic parameters ,anxiety, sedation score , and pain during block and surgery, satisfaction of surgeon were assessed. . At the preoperative visit verbal pain score (VPS) of 10 (0 = no pain and 10 = worst pain imaginable) and verbal anxiety score (VAS) ranging from 0 to 10 (0= completely calm, 10 = the worst possible anxiety) were explained to patients. Then a 20 gauge cannula was inserted into one of the two hands. Patients were monitored with electrocardiogram, noninvasive measurement of blood pressure, and pulse oximetry (SPO2). Retrobulbar nerve block was performed by the same ophthalmic surgeon who was unaware of group allocation with 1.5 ml of solution that prepared by nurse( lidocaine 2%and 0.5 ml bupivacaine) via the percutaneous route with a 25 G, 38 mm Atkinson needle (John Weiss & Son Limited, Milton Keynes,England), at inferotemporal site. No patient received an additional facial nerve block. The investigators assessed the pain immediately after block and surgery. Anxiety score and pain score was recorded in each patient before premedication (T1), ninety minutes after premedication, on arrival in the operating room (T2), one minute after retrobulbar block placement (T3)during the operation period) (T4) and postoperatively before discharging the patient from the recovery room (T5) .At the end of surgery, the patients were asked about average level of their anxiety and pain during the operation period according to the VAS and VPS explained to them before premedication.'. The surgeon was also asked to verbally rate their level of satisfaction according to three degree scale as "very bad, , moderate, good after the operation. The sedation level of patients during performance of block was assessed as Sedation scores were obtained on a 3 point scale with 0 =movements of the head, arms and trunk ,1 =slightly movement of arms,2=slightly change in face,3=complete calm. If sedation was inadequate, fentanyl could be given 0.5microgram/kg as needed.

ELIGIBILITY:
Inclusion Criteria:

* patients who were aged 25 years or older, American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Patients with ASA status IV
* history of hepatic or renal disease, confusion, dementia
* communication difficulty resulting from deafness or language barrier
* chronic use of narcotics, barbiturates or psychotropic medications
* history of allergy or contraindications to any of the study drugs
* visual impairment of the non operative eye
* weight < 40 kg or > 100 kg

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
pain will be assessed by verbal pain score (VPS) of 10 (0 = no pain and 10 = worst pain imaginable) | one minute after retrobulbar block placement
pain will be assessed by verbal pain score (VPS) of 10 (0 = no pain and 10 = worst pain imaginable) | At the end of surgery the patients were asked about average level of their pain during the operation period according to the VPS explained to them before premedication)
pain will be assessed by verbal pain score (VPS) of 10 (0 = no pain and 10 = worst pain imaginable) | postoperatively before discharging the patient from the recovery room
anxiety will be assessed by verbal anxiety score (VAS) of 10 (0 = completely calm and 10 = the worst possible anxiety) | At the end of surgery the patients were asked about average level of their pain during the operation period according to the VPS explained to them before premedication)
anxiety will be assessed by verbal anxiety score (VAS) of 10 (0 = completely calm and 10 = the worst possible anxiety) | one minute after retrobulbar block placement
anxiety will be assessed by verbal anxiety score (VAS) of 10 (0 = completely calm and 10 = the worst possible anxiety) | postoperatively before discharging the patient from the recovery room

SECONDARY OUTCOMES:
mean arterial blood pressure will be assessed by noninvasive automatic blood pressure measurement | before premedication
mean arterial blood pressure will be assessed by noninvasive automatic blood pressure measurement | ninety minutes after premedication, on arrival in the operating room
mean arterial blood pressure will be assessed by noninvasive automatic blood pressure measurement | one minute after retrobulbar block placement
mean arterial blood pressure will be assessed by noninvasive automatic blood pressure measurement | during the operation period(five minutes after beginning of surgery
mean arterial blood pressure will be assessed by noninvasive automatic blood pressure measurement | postoperatively before discharge the patient from the recovery room
heart rate will be assessed by echocardiogram monitoring | before premedication
heart rate will be assessed by echocardiogram monitoring | ninety minutes after premedication, on arrival in the operating room
heart rate will be assessed by echocardiogram monitoring | one minute after retrobulbar block placement
heart rate will be assessed by echocardiogram monitoring | during the operation period(five minutes after beginning of surgery
heart rate will be assessed by echocardiogram monitoring | postoperatively before discharge the patient from the recovery room
satisfaction of surgeon according to three degree scale as very bad, moderate, good will be assessed | one minute after retrobulbar block placement
satisfaction of surgeon according to three degree scale as very bad, moderate, good will be assessed | at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin university of medical science, Qazvin, Qazvin Province, Iran